CLINICAL TRIAL: NCT07070453
Title: Effect of Photodynamic Therapy as an Adjunct to Non-Surgical Treatment of Periodontitis
Acronym: PerioFPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Egas Moniz - Cooperativa de Ensino Superior, CRL (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: aPDT FPS; CiiEM Investiga (Other Grant/Funding Number: Egas Moniz School of Science and Health)
Record Dates: First submitted 2025-01-24; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Periodontitis
Keywords: periodontitis; antimicrobial photodinamic therapy
MeSH Terms: conditions — Periodontitis | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-surgical periodontal treatment (Active Comparator): Conventional non-surgical treatment - scaling and root planing
  Interventions: Procedure: Non-surgical periodontal treatment
- Antimicrobial photodynamic therapy (Experimental): Scaling and root planing + aPDT (antimicrobial photodynamic therapy)
  Interventions: Procedure: Scaling and root planing + aPDT

INTERVENTIONS:
Procedure: Non-surgical periodontal treatment — Removal of deposits above and below the gum line using hand or ultrasonic tools and thorough smoothing of root surfaces to discourage re-accumulation of bacteria.
  Arms: Non-surgical periodontal treatment
Procedure: Scaling and root planing + aPDT — Non-invasive treatment that uses a combination of a light-sensitive compound (photosensitizer), specific light, and oxygen to generate reactive oxygen species (ROS) that kill bacteria.
  Arms: Antimicrobial photodynamic therapy

SUMMARY:
Photodynamic therapy (PDT) is an innovative technique that utilizes light-activated agents, known as photosensitizers, to produce reactive oxygen species capable of targeting and eliminating pathogens. This therapeutic approach has been explored in a variety of medical fields due to its versatility and minimal invasiveness. In the context of periodontal diseases, PDT has emerged as a promising adjunctive treatment in the non-surgical management of periodontitis. Periodontitis, a chronic inflammatory disease caused by the accumulation of pathogenic bacteria in the subgingival environment, is often treated with mechanical debridement, including scaling and root planing (SRP). However, these conventional methods may not always achieve complete bacterial eradication. PDT, when used in conjunction with SRP, has the potential to significantly enhance bacterial elimination. The use of photosensitizers, activated by specific wavelengths of light, leads to the generation of singlet oxygen, which can effectively kill a broad spectrum of periodontal pathogens, including those resistant to antibiotics. As an adjunctive therapy, PDT can improve the clinical outcomes of non-surgical periodontitis treatment by reducing bacterial load, promoting tissue healing, and potentially decreasing the need for more invasive procedures. The ability of PDT to target bacteria without harming surrounding tissues makes it an attractive option for patients who require a non-invasive treatment approach. In conclusion, photodynamic therapy is a valuable addition to periodontal treatment regimens, offering enhanced bacterial reduction and improved therapeutic outcomes in the management of periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older with periodontitis diagnosed according to EFP/APA 2018 criteria and with at least 10 teeth in the mouth.

Exclusion Criteria:

* Periodontal treatment in the previous six months; use of antibiotics, NSAIDs or immunosuppressants in the previous six months; acute oral infection; pregnant or breastfeeding women; teeth with grade III mobility; pockets with PD > 10 mm; use of antimicrobial mouthwash in the previous two months; patients with diabetes mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Microbiology outcome | From enrollment to the end of treatment at 3 months.
  Changes in the microbiome collected from periodontal pockets sequencing 16S ribosomal RNA gene

SECONDARY OUTCOMES:
Clinical outcome | From enrollment to the end of treatment at 3 months.
  Probing depth, measuring in millimeters the distance from the gingival margin to the base of a sulcus or periodontal pocket, using a periodontal probe.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Dr. Alves, phd, Principal Investigator — Egas Moniz School of Science and Health
Locations (1):
- Egas Moniz School of Health and Science, Almada, Monte Da Caparica, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: LED site — https://www.bredent-implants.com/products-solutions/regeneration/helbo/